CLINICAL TRIAL: NCT05156879
Title: Low Dose of Aspirin for the Management of Endometriosis-associated Pelvic Pain: a Randomized, Open, Controlled Trial
Brief Title: Aspirin for the Management of Endometriosis-associated Pelvic Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20210267-R
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Aspirin; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Aspirin Enteric-coated Tablets，75mg/day，24 weeks
  Interventions: Drug: Aspirin
- Drospirenone ethinyl estradiol (Active Comparator): Drospirenone ethinyl estradiol，one tablet/day for 21 consecutive days, 28 days as a cycle of use，24 weeks
  Interventions: Drug: Drospirenone ethinyl estradiol

INTERVENTIONS:
Drug: Aspirin — 75mg, one time/day
  Arms: Aspirin
Drug: Drospirenone ethinyl estradiol — 1 table/day, 21 consecutive days, 28 days as a cycle of use
  Arms: Drospirenone ethinyl estradiol

SUMMARY:
Endometriosis-associated pelvic pain (EAPP) is common in endometriosis and pain control is an important goal of long-term management. Non-steroidal anti-inflammatory drugs and oral contraception are the two first line therapies for endometriosis. High quality study about aspirin for the EAPP is absent. In this study, the investigators hypothesis that aspirin is effective in controlling EAPP. A randomized, open, and controlled study will be implemented. "participants with EAPP with visual Analogue Scale(VAS）>30 mm will be included and low dose aspirin（75mg/day） be prescribed. Yasmin(Drospirenone ethinyl estradiol tablet) will be used as positive control. The primary efficacy end points is the reduction of the pain score of EAPP at 24th week assessed with VAS score. Pelvic examination, sonography and blood test will be to performed to evaluate the lesion and coagulation function. The adverse event and medication compliance will be investigated. The aim of this study is to explore the efficacy and safety of low dose aspirin therapy in management of EAPP. This study will provide new options for the long-term management of endometriosis, which will help reduce the medical cost of endometriosis.

DETAILED DESCRIPTION:
Endometriosis-associated pelvic pain (EAPP) is common in endometriosis and pain control is an important goal of long-term management. Non-steroidal anti-inflammatory drugs and oral contraception are the two first line therapies for endometriosis.However, there is currently a lack of high-quality clinical studies of nonsteroidal anti-inflammatory analgesic in controlling EAPP. The aim of this study is to explore the efficacy and safety of low dose aspirin therapy in management of EAPP. In this study, the investigators hypothesis that aspirin is effective in controlling EAPP. A randomized, open, and controlled study will be implemented. Subjects were recruited in strict accordance the inclusion and exclusion criteria at the outpatient clinic. Patients with EAPP with visual Analogue Scale(VAS:0-100mm）>30mm will be included. Eligible subjects were randomized according to a computer-generated randomization schedule to to receive aspirin（75mg/day）or Yasmin(Drospirenone ethinyl estradiol tablet) in a ratio of 1:1. Specific doctors will be designated for the disease diagnosis and ultrasonic examination.The investigators were guided by EAPP pain score and drug use management. The primary efficacy end points is the reduction of the pain score of EAPP at 24th week assessed with VAS score. Pelvic examination, sonography and blood test will be to performed to evaluate the lesion and coagulation function. The specification of the CONSORT case report system will be implemented. Sample size assessment according equivalence study.Follow-up and loss cases were strictly controlled. A two-sided test will performed with beta=0.80 and αlpha=0.025. The expected loss rate is calculated at 15%. 220 cases will be enrolled with 110 cases in each group. The study will be accepted regular monitoring and inspection.

ELIGIBILITY:
Inclusion Criteria:

* Dysmenorrhea or non-cyclical pelvic pain lasts for more than 3 months, and the VAS pain score is larger than 30mm
* diagnosed as endometriosis
* Willing to participate in clinical trials and sign informed consent

Exclusion Criteria:

* Those who have a clear surgical treatment plan due to various diseases within 6 months
* Suspected or suffering from malignant tumor
* Hemoglobin less than 8g/dl
* women with contraindications to the use of aspirin or oral contraceptives
* with other painful disease other than endometriosis
* Active bleeding from other areas or undiagnosed abnormal vaginal bleeding
* drug adminstration within 3 months including oral contraceptives, dienogest, Mirena or GnRH-a preparations, analgesics/Chinese medicines or proprietary Chinese medicines, etc.
* Pregnancy status or breastfeeding
* Any disease or symptom that may affect the implementation of the study or the interpretation of the results
* Participate in other clinical trials at the same time

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 220 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
visual Analogue Scale | baseline , 12 weeks after treatment , and 24 weeks of treatment
  a scale with 0-100 mm values, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Tenderness | baseline , 12 weeks of treatment , and 24 weeks of treatment
  Tenderness during pelvic examination from 1 to 4,higher scores mean a worse outcome
size of endometrioid lesions | baseline , 12 weeks of treatment , and 24 weeks of treatment
  endometrioid lesions detected by sonorgraphy
C reactive protein | baseline , 12 weeks of treatment , and 24 weeks of treatment
  a biomarker of inflammation
carbohydrate antigen 125 | baseline , 12 weeks of treatment , and 24 weeks of treatment
  a biomarker of endometriosis
platelets counts | baseline , 12 weeks of treatment , and 24 weeks of treatment
  associated with inflammation and wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Zhengyun Chen, Master, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No